CLINICAL TRIAL: NCT04875494
Title: Physical Exercise and Self-esteem: a Randomized Controlled Trial in Domestic Violence Victims
Brief Title: Effects of Physical Exercise Versus Group Therapy on Self-esteem Among Domestic Violence Victims
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Principal Investigator, Fabien Legrand, Clinical Professor, Université de Reims Champagne-Ardenne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DDCSPP
Record Dates: First submitted 2021-04-21; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Domestic Violence
MeSH Terms: interventions — Counseling; Exercise

STUDY DESIGN:
Intervention Model Description: Three independant groups including two intervention groups (Physical Exercise vs. Group Therapy) and one control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical Exercise (Experimental)
  Interventions: Behavioral: Physical Exercise
- Counseling/support group therapy (Active Comparator)
  Interventions: Behavioral: Counseling/support group therapy
- Control (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Counseling/support group therapy — 6 weeks of counseling group therapy; 2 sessions of 30 min each week, with a psychologist and two former victims
  Arms: Counseling/support group therapy
Behavioral: Physical Exercise — 6 weeks of physical exercise training; 2 sessions of 30 min each week, with an instructor
  Arms: Physical Exercise

SUMMARY:
The current study is a randomized controlled trial comparing the effects of 6 weeks of physical exercise training versus group therapy on self-esteem as well as on the various subdomains of physical self-esteem among women who have experienced domestic violence within the last two months at the time of data collection

DETAILED DESCRIPTION:
The present study design includes three arms (two intervention arms): Physical Exercise (Group A), Counseling/Support Group (Group B), and No Intervention (Control, Group C). Random allocation to each group was done in a 1:1:1 ratio at the end of an initial telephone interview by one of the authors. A permutated block design with a block size of three was used. For each participant in Groups A and B, the assigned intervention was started the week following the initial interview, and lasted 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* having experienced domestic violence at some time in the past 2 months

Exclusion Criteria:

* not being physically active on a regular basis (less than 20 min of moderate-vigorous physical activity per day during the last year)
* absence of medical contraindication to exercise

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Change score for each of the physical and global self esteem subscales from the Inventaire du Soi Physique (ISP-25). This instrument has 25 items each with a 6-point Likert response scale. Higher scores indicate greater self-esteem (physical or global) | baseline (pre-): the day before intervention implementation; post-study: the day following cessation of intervention, 6 weeks from baseline
  magnitude of change in global and physical self-esteem from pre- to post-study. Minimum = -150; Maximum = +150

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie CAILLIES, PhD, Study Director — Université de Reims Champagne-Ardenne
Locations (1):
- CIDFF-51, Châlons-en-Champagne, France

IPD SHARING:
Plan to Share IPD: No